CLINICAL TRIAL: NCT00443885
Title: Resistance Rates and Mechanisms of Resistance to Imipenem and Meropenem at UPMC to Problematic Gram-negative Organisms
Brief Title: Resistance Rates and Mechanisms of Resistance to Imipenem and Meropenem at UPMC
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Brian Potoski, Pharm D, University of Pittsburgh
Other Study IDs: PRO07020078
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Gram Negative Organism
Keywords: meropenem; imipenem; gram negative organism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The isolate samples will be collected over a period of one year once IRB approval has been obtained. These isolates were collected as part of the patient's clinical care and once all clinical testing is complete, all isolates will be discarded. The honest broker of our area will collect the isolates and deidentify all information once all clinical testing is complete. The isolates will be obtained from the microbiology lab.

DETAILED DESCRIPTION:
The study will collect two hundred pseudomonas and 20 acinetobacter baumanti consecutive bacterial isolates from microbiology. These isolates are collected as part of the patient's clinical care and are discarded once all clinical testing is complete. The honest broker will obtain these samples after all clinical testing is complete. All isolates will be deidentified. These isolates will be tested using standardized susceptibility methods for meropenem and imipenem. The activity of doripenem, a carbapenem currently being studied, and arbekacin an aminoglycoside, will also be tested. The honest broker will also collect limited patient data including underlying condition, presence of a solid organ transplant, ward location, and antibiotic history over the three months prior to organism isolation. For resistant isolates found, analytical and molecular techniques will be performed to determine the mechanisms of resistance and whether resistant isolates are coming from a single source/being transmitted from person to person.

ELIGIBILITY:
Inclusion Criteria:

* Samples" for the purpose of this study are Gram negative bacteria in a Petri dish of growth media.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: gram negative bacteria
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2007-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
dead or alive | end of study
  health status

CONTACTS AND LOCATIONS:
Overall Officials: Brian Potoski, Pharm D, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania